CLINICAL TRIAL: NCT03523312
Title: Maximal Ablative Irradiation Because of Encasement (MAIBE) for Patients With Potentially Resectable Locally Advanced Pancreatic Cancer
Brief Title: Use of High-dose Radiation Therapy Plus Chemotherapy to Improve the Likelihood of Surgical Treatment in Patients With Locally Advanced Pancreatic Cancer
Acronym: MAIBE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-090
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: Ablative Irradiation; 18-090
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: This phase II trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HFA-IMRT (Experimental): Eligible patients will receive HFA-IMRT to a total dose of 67.5 Gy in 15 fractions or 75Gy in 25 fractions to areas of gross tumor with concurrent capecitabine. Cross-sectional imaging will be repeated 4-6 weeks after the end of CRT to assess for resectability.
  Interventions: Radiation: Hypofractionated ablative IMRT (HFA-IMRT); Drug: capecitabine

INTERVENTIONS:
Radiation: Hypofractionated ablative IMRT (HFA-IMRT) — total dose of 67.5 Gy in 15 fractions or 75Gy in 25 fractions
Drug: capecitabine — Oral capecitabine at 825 mg/m2 BID on the days of RT. 5 Fluorouracil (5FU) at 250mg/m2/day, 7 days per week by a continuous IV infusion via an outpatient infusion pump) may be used instead at the discretion of the treating physician.

SUMMARY:
This study is being done to test whether receiving a dose of radiation that is higher than the standard dose, in combination with chemotherapy, improves the chance of becoming a candidate for surgery and improves the chance of extending the patient's life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytopathologically confirmed adenocarcinoma of the pancreas.
* Locally advanced, unresectable pancreatic cancer defined on post-induction chemotherapy CT as having tumor involvement of >180° (> 50%) of the circumference of the superior mesenteric artery (SMA) or celiac axis, unreconstructable superior mesenteric vein (SMV) or PV involvement.
* No evidence of distant metastasis either prior to or after induction chemotherapy.
* Completion of at least 3 months of standard induction chemotherapy for LAPC, which may include FOLFIRINOX or gemcitabine and nab-paclitaxel, within 6 weeks of enrollment.
* For patients currently receiving investigational agents, a washout of at least 2 weeks or 5 half-lives of experimental agent are required prior to the start of RT.
* Age ≥18 years.
* KPS 70-100.
* Patients must have acceptable organ and marrow function as defined below:

  * Leukocytes >3,000/µL
  * Absolute neutrophil count >1,500/µL
  * Platelets >75,000/µL
  * Total bilirubin Within 2 x upper limit of normal
  * AST (SGOT)/ALT (SGPT) <2.5 x institutional upper limit of normal Creatinine Within 1.5 x upper limit of normal, OR Creatinine clearance >60 mL/min for patients with creatinine levels above institutional normal
* Any systemic therapy associated toxicity should be Grade 1 or less
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have borderline resectable disease using NCCN definition.
* Patients who have had prior abdominal radiotherapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Patients who are not surgical candidates due to medical co-morbidities.
* Patients in whom iodine contrast is contraindicated.
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 4 weeks after the study are excluded. This applies to any woman who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months, or women on hormone replacement therapy with serum FSH levels greater than 35 mIU/mL. A negative serum pregnancy test must be obtained within 14 days prior to the start of study therapy in all women of child-bearing potential. Male subjects must also agree to use effective contraception for the same period as above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who undergo definitive surgery | 2 years
  The proportion of patients who undergo definitive surgery will be used to evaluate efficacy of HFA-IMRT in improving rates of resectability as compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Reyngold, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm